CLINICAL TRIAL: NCT06201611
Title: A 3-arm, Open-label, Stratified Randomized Controlled Trial With Blinded End-point Assessment to EValuate A Nitric oxidE Generator (Nebivolol) as a diSease Modifying mediCatioN in Diabetic Peripheral Neuropathy
Brief Title: Evaluating a Nitric Oxide Generator, Nebivolol as a Disease Modifier in Patients With Diabetic Neuropathy.
Acronym: EVANESCENT-DPN
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: St. John's Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IEC/1/1218/2023
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Neuropathy Peripheral
MeSH Terms: interventions — epalrestat

STUDY DESIGN:
Intervention Model Description: We will use a 3 center, 3-arm, parallel group, open label, stratified randomized controlled trial design with a 1:1:1 allocation ratio and blinding of outcome assessors.
Who Masked: Outcomes Assessor
Masking Description: Trained outcomes assessor unaware of the treatment arm to which the patient has been allocated to will perform all outcomes assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Nebivolol+ Standard care arm (Experimental): This arm will receive tablet Nebivolol 2.5 mg OD uptitrated at 2 weeks to 5 mg and at 4 weeks if well tolerated to 10 mg/day which the participant will continue upto week 24
  Interventions: Drug: Nebivolol+ Standard care arm
- Epalrestat + Alpha Lipoic Acid +Standard care (Active Comparator): This arm will receive tablet Epalrestat -150mg OD+ cap Alpha Lipoic Acid 600mg OD for 24 weeks.
  Interventions: Drug: Epalrestat + Alpha Lipoic Acid +Standard care
- Standard care alone (Active Comparator): Patients in this arm will receive standard care as judged by their treating physicians which is generally pain modifying treatment.
  Interventions: Drug: Standard care alone

INTERVENTIONS:
Drug: Nebivolol+ Standard care arm — This arm will receive tablet Nebivolol 2.5 mg OD uptitrated at 2 weeks to 5 mg and at 4 weeks if well tolerated to 10 mg/day which the participant will continue upto week 24
  Arms: Nebivolol+ Standard care arm
Drug: Epalrestat + Alpha Lipoic Acid +Standard care — This arm will receive tablet Epalrestat -150mg OD+ cap Alpha Lipoic Acid 600mg OD for 24 weeks.
  Arms: Epalrestat + Alpha Lipoic Acid +Standard care
Drug: Standard care alone — Patients in this arm will receive standard care as judged by their treating physicians which is generally pain modifying treatment.
  Arms: Standard care alone

SUMMARY:
The goal of this clinical trial is to test in patients with diabetic neuropathy,

* Can Nevibolol at a dose of 2.5 mg- 10 mg compared with standard pain modulating treatment conserve the mean nerve action potential amplitude (sural and tibial nerves) at 24 weeks follow- up.
* Can Nevibolol at a dose of 2.5 mg- 10 mg compared with a combination of Alpha Lipoic Acid (600 mg/day)+EPALRESTAT (150 mg/day) conserve the mean nerve action potential amplitude (sural and tibial nerves) at 24 weeks follow- up

  * All potential participants will undergo screening- about 10 ml of blood will be drawn to perform the following assesments at screening- HbA1c, FBS,Vit B12, TSH, fT4.
  * Baseline assessments conducting a nerve conduction study, quality of life assesment using Eq-5D-5L and NRS pain score.
  * 20% of patients (24 patients) will undergo Sudoscan, Corneal confocal microscopy and a skin biopsy for assessing IENFD (Intra Epidermal Nerve Fibre Density).
  * 15th day, 1 month and 3rd month followup for evaluating patients status and medication adherance.
  * 6th month followup for evaluating patients status and medication adherance.

Researchers will compare Nebivolol against combination of Epalrestat+Alpha Lipoic Acid against standard pain modulating treatment to evaluate their diseaes modifying effect as reflected by nerve conduction study parameters.

DETAILED DESCRIPTION:
A 3 centre, 3-arm, parallel group, open label, stratified randomized controlled trial design is used with a 1:1:1 allocation ratio and blinding of outcome assessors.

Primary Objectives:

1. To evaluate the efficacy of Tab. Nebivolol 10 mg/ day (or maximally tolerated dose) compared to standard care (pain modulators alone) on mean nerve action potential at week 24.
2. To evaluate the efficacy of Tab. Nebivolol 10 mg/day (or maximally tolerated dose) compared to a combination of lipoic acid 600 mg/d plus epalrestat 150 mg/day at week 24 on mean nerve action potential at week 24.

Secondary Objectives: 1. To compare the intra-epidermal nerve fibre density (IENFD), high-sensitivity C-reactive protein (hsCRP) and quantify GAP-43 (neuromodulin) in a randomly selected sample (stratified by sex and baseline disease severity) of 20% patients from each from the 3 arms pre and post intervention: corneal nerve fiber length and density using confocal microscopy in all patients in the 3 arms at week 24.

2. To compare the electrical conductance (mean µSiemens) using Sudoscan between the nebivolol arm versus standard care alone and the nebivolol arm versus alpha-lipoic acid plus epalrestat arm at week 24.

3.To compare mean hsCRP levels in a randomly selected sample of 20% of patients between the 3 arms at 6 months and change in mean hsCRP levels from baseline to 6 months in the intervention arm.

4) To compare mean GAP-43 levels in a randomly selected sample of 20% of patients.

5) To compare mean intra-epidermal nerve fiber density (IENFD) in a randomly selected sample of 20% of patients.

6)To compare corneal nerve fiber length and density in a randomly selected sample of 20% of patients.

7) Electrical conductance (mean µSiemens) using Sudoscan between the nebivolol arm versus standard care alone and the nebivolol arm versus alpha-lipoic acid plus epalrestat arm at week 24.

8) Mean nerve conduction velocity - nebivolol versus standard care and nebivolol versus alpha-lipoic acid+epalrestat arms at week 24.

9) Compare general quality of life measured using the EQ-5D-5L questionnaire at week 24.

10) Cost-effectiveness analysis between the three treatment arms with nerve conduction study parameters and numerical pain rating scores as outcome measures at week 24.

Patients will be randomized into three of the following arms- Arm 1 - Tab. Nebivolol 2.5 mg/day from baseline to week 2, up-titrated to 5 mg/day at week 2 and from 5 mg/ day to 10 mg/day from week 4 to week 24 after an ECG at week 4 plus standard care pain modulating drugs.

Arm 2 - Cap. Alpha-Lipoic Acid 600 mg/ day plus Tab. Epalrestat 150 mg/day from baseline to week 24 plus standard care pain modulating drugs.

Arm 3 - Standard pain modulating treatments per physician's discretion. This will likely be a monotherapy or combinations of pregabalin, duloxetine or amitriptyline.

Only patients with stable glycemic control for the past 3 months will be enrolled. During screening if patients has uncontrolled diabetes, the doses of the diabetes treatments will be optimized, add-on treatments will be commenced and if needed medications for risk factor control such as statins and anti-hypertensives will be added on. All patients will receive dietary counselling for medical nutrition therapy (MNT) and guideline-based exercise regimen advised. Glycemic control and adherence to all standard care treatments will be periodically assessed at follow-ups and encouraged. Rescue Medications - Tab. Paracetamol 1 gram up to 4 grams over a 24 hour period will be added in cases of intractable pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged >= 18 years diagnosed with diabetes mellitus, of a duration of <= 5 years since their diagnosis
2. HbA1c < 9 at enrolment with stable glycemic control for the last three months
3. Neuropathy meeting the following 'Toronto criteria' (8) - (a) abnormal nerve conduction study* based on age-matched controls at the site and - (b) a symptom or sign of neuropathy defined as one of either a diabetic neuropathy symptom score of >= 1/4 Or neuropathy disability score of >= 3/10 (9).

   * Abnormal NCS defined as one or more abnormal Z score in two or more nerves, based on sural nerve amplitude (antidromic stimulation), tibial and peroneal NCV, tibial amplitude, increased F-wave minimum latency (F-min), and absent F-waves (only considered abnormal in tibial nerve)

Exclusion Criteria:

1. Absolute contra-indications for nebivolol - sick-sinus syndrome, sinus bradycardia with a resting heart rate < 50/ minute, second or third degree AV-nodal blocks fascicular blocks, severe asthma or COPD and acute heart failure
2. Patients with a compelling indication for a non-dihydropyridine calcium channel blocker (CCB)
3. Patients with compelling need for another beta-blocker in the judgement of the treating team

Patients who have undergone major amputations of the lower limbs or are posted for the same.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
The mean nerve action potential amplitude (sural and tibial nerves) between Arm 1 and Arm 3 at 24 weeks follow-up. | Baseline and 24 weeks
  As part of nerve conduction study, the mean nerve action potential amplitude (sural and tibial nerves) will be compared between Arm 1 and Arm 3 at 24 weeks follow-up.

SECONDARY OUTCOMES:
The proportion of patients who progress to develop severe neuropathy | Baseline and 24 weeks
  To compare -
  1. The proportion of patients who progress to severe neuropathy at week 24 follow-up.
  2. The proportion of patients having a pain numerical rating scale(NRS) score & between Nebivolol, lipoic acid+epalrestat and standard care arms at weeks 4 and 12.
  3. Quantifying the intra-epidermal nerve fibre density (IENFD), high-sensitivity C-reactive protein (hsCRP) levels and GAP-43 (neuromodulin) in a randomly selected sample (stratified by sex and baseline disease severity) of 20% patients each from the 3 arms pre and post-intervention and corneal nerve fibre length and density in all patients in the 3 arms at week 24.

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - St John's Medical College Hospital, Bangalore, Karnataka
  - St John's Research Institute, Bangalore, Karntakaka

IPD SHARING:
Plan to Share IPD: Yes
The Sponsors St John's Research Institute will be the primary custodians of the data. The anonymized identified data will be shared on an open access database 3 years after declaring the database lock. After publishing the primary results , interested researchers can approach the sponsors with a research question and a protocol. This will be evaluated by the sponsors and if found meritorious the sponsors may share the data with the investigators who have applied
Supporting Information: Study Protocol, ICF
Time Frame: 3 years after database lock indefinitely.